CLINICAL TRIAL: NCT02445521
Title: Testing of Four Home Phenylalanine Monitoring Prototype Devices Using Whole Blood From Normal and PKU Subjects
Brief Title: Testing of Four Home Phenylalanine Monitoring Prototype Devices
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: National PKU Alliance (Unknown)
Responsible Party: Principal Investigator, Rani Singh, Professor, Emory University
Other Study IDs: IRB00079788
Record Dates: First submitted 2015-05-13; First posted 2015-05-15 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-12

CONDITIONS: Phenylketonurias
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Whole blood and plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (5):
- PKU (low phe-level): A subject diagnosed with phenylketonuria (PKU) with low phenylalanine levels, defined as 1-5 mg/dL
- PKU (mid phe-level): A subject diagnosed with phenylketonuria (PKU) with middle phenylalanine levels, defined as 6-10 mg/dL
- PKU (high mid phe-level): A subject diagnosed with phenylketonuria (PKU) with high middle phenylalanine levels, defined as 11-15 mg/dL
- PKU (high phe-level): A subject diagnosed with phenylketonuria (PKU) with high phenylalanine levels, defined as 16-20+ mg/dL
- Control: A normal subject without phenylketonuria (PKU)

SUMMARY:
The objective of this study is to test four home phenylalanine monitoring prototype devices, selected out of a pool of candidates by the National PKU Alliance Scientific Committee.

DETAILED DESCRIPTION:
A real time, point-of-care and home phenylalanine monitoring system would provide patients with quick results and feedback. Home monitoring devices' phenylalanine measurements will be compared to the current gold-standard measurement of phenylalanine (plasma concentration) in four subjects with PKU and one control subject. The study will enroll subjects with different baseline phenylalanine concentrations (i.e., patients with poor to good metabolic control, assessed by comparing current phenylalanine concentrations to established treatment ranges).

For each prototype device, three separate measurements of phenylalanine per subject will be performed. Three prototype devices require whole blood, thus 1 teaspoon (approximately 4mL) of whole blood will be collected through venipuncture and blood spots will be used to conduct tests. One prototype requires capillary blood to be collected through a fingerstick, and will require three blood spots from the stick. A single plasma amino acid analysis for each participant will also be performed using leftover whole blood from the 4mL blood draw through quantitative ion exchange chromatography, reported as micromoles/L.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of PKU or hyperphenylalaninemia (PKU group)
* any age
* in good health (PKU and control group)

Exclusion Criteria:

* pregnant
* have any medical comorbidities
* considered unfit for participation by the principal investigator

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Control will be recruited by distributing an email to all staff on the Emory Genetics Clinic listserv to solicit a volunteer to provide 4ml of whole blood only. Respondents who are within two years of age and the same gender of at least one of the PKU subjects will be considered eligible. Remaining subjects will be recruited through Emory Genetics Clinic and possibly through the Emory Metabolic Nutrition Program's Annual Metabolic Camp.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2015-05; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Intra-variability of the four devices, assessed by phenylalanine values | Day 1
  Phenylalanine values for each of the three runs on each device for the same individual will be compared. Each PKU subject will be assessed separately to assess the reliability of each device since the subjects will have a range of phenylalanine concentrations.

SECONDARY OUTCOMES:
Inter-variability of the four devices, assessed by average phenylalanine concentrations | Day 1
  Average phenylalanine values measured by the four tests of each device in each subject will be calculated. Mean concentrations for each device will be compared to the control (gold standard measure of plasma phenylalanine).

CONTACTS AND LOCATIONS:
Overall Officials: Rani H Singh, PhD, RD, LD, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Children's Healthcare of Atlanta (CHOA), Atlanta, Georgia
  - Emory University Hospital - Atlanta Clinical and Translational Science Institute (ACTSI), Atlanta, Georgia
  - Emory University Genetics Clinic, Decatur, Georgia